CLINICAL TRIAL: NCT07157618
Title: Development and Clinical Application of Deep Learning-Based Prospective Pathology Foundation Models
Brief Title: Prospective Pathology Foundation Models
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-403
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pancancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples Without DNA: Samples retained, with no potential for DNA extraction from any retained samples (e.g., fixed tissue, plasma)

GROUPS / COHORTS (3):
- QFSH external validation dataset: 1000 slides from 1000 eligible individuals were obtained in the Qianfoshan Hospital (QFSH, Jinan, China) between January 2020 and July 2025, which was used to validate the pathology foundation models.
- Prospective validation dataset: We conducted a prospective validation study to compare the diagnostic performance among pathologists, our pathology foundation model, and pathologist-with-AI-assisted diagnosis. This study was initiated on August 28, 2025 at Nanfang Hospital, Southern Medical University (NFHSMU).
- Randomized controlled trial: We conducted a prospective randomized controlled trial to compare the diagnostic performance among pathologists, the pathology foundation model, and pathologist-with-model-assisted diagnosis at Nanfang Hospital of Southern Medical University (NFHSMU).The trial commenced data collection on August 28, 2025 to establish the NFHSMU randomized controlled trial dataset. Following quality control, the slides were randomly allocated (1:1:1 ratio) into three groups:Model-only group/Pathologist-only group/Model-assisted pathologist group.

SUMMARY:
Histopathology remains the gold standard for disease diagnosis, yet faces challenges including pathologist shortages and diagnostic model limitations. This underscores the critical need to develop deep learning-based pathology foundation models integrating prospective imaging and clinical data. Such models would enhance diagnostic accuracy and efficiency, enabling tumor grading, histo-molecular classification, and intelligent chemotherapy guidance - ultimately optimizing clinical workflows. However, a critical gap remains: the absence of prospectively validated, pan-disease pathology foundation models. Developing clinically validated models is therefore imperative.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old.
2. Patients with complete pathological slides and clinical information.

Exclusion Criteria:

1.Patients with missing data or specimens not meeting quality control requirements for analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria comprised patients aged 18-75 years with definitive pathological diagnoses. All cases were prospectively collected from Nanfang Hospital, Southern Medical University (NFHSMU) .
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Area under ROC curve (AUC) | Diagnostic evaluation will be performed within 1 week when the WSIs are obtained
  Area under the curve

SECONDARY OUTCOMES:
Specificity | Diagnostic evaluation will be performed within 1 week when the WSIs are obtained
  The true negative rate (TNR) of the diagnostic platform, which is the ratio between the number of negative individuals correctly categorized by platform and the total number of actual negative individuals (%).
Sensitivity | Diagnostic evaluation will be performed within 1 week when the WSIs are obtained
  The true positive rate (TPR) of the diagnostic platform, which is the ratio between the number of positive individuals correctly categorized by platform and the total number of actual positive individuals (%).

CONTACTS AND LOCATIONS:
Overall Officials: Li Liang, Study Director — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Qianfoshan Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No
Requests for the data collected and analyzed in this study will be considered if the application is in line with public benefits and the applicant is willing to sign a data access agreement. Contact can be through the corresponding author.